CLINICAL TRIAL: NCT04240652
Title: The Diabetic Retinopathy Screening, Prevention and Control Program
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Ruijin-20191231
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — DNA, Serum and plasma are retained
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with fundus photography: Subjects diagnosed with diabetes or not who have fundus images from MMCs and other medical institutes.

SUMMARY:
The greatest harm of diabetes is various acute and chronic complications, especially diabetic retinopathy(DR), leading to extremely high rates of disability and blindness. Early screening, early diagnosis, and early treatment are the keys to maintaining vision in patients with DR. However, compared with the high prevalence of diabetes in China, the DR screening ability is relatively inadequate. To change this situation, deep learning(DL), a form of artificial intelligence (AI), might be a potential effective method to solve this dilemma.

DETAILED DESCRIPTION:
The greatest harm of diabetes is various acute and chronic complications, especially DR, leading to extremely high rates of disability and blindness. However, if the fundus examination is carried out regularly in the early stages of onset, the risk of blindness can be significantly reduced. Therefore, early screening, early diagnosis, and early treatment are the keys to maintaining vision in patients with DR. However, compared with the high prevalence of diabetes in China, the DR screening ability is relatively inadequate.

The Diabetic Retinopathy Screening and Prevention Program is a branch project of MMC. Its purpose is to carry out an efficient workflow for early detecting, timely managing of DR, and to establish a referral system for implementing treatment and the long-term follow-up of DR by means of DL. First, In order to improve its sensitivity and specificity, more participants are involved in other medical institutes besides MMCs, then we can effectively explore the prevalance of DR in China and helps to early screening, prevention, treatment and referal process of DR. Secend, we collect participants' serum, plasma,DNA, several medical stastistics and life styles to explore genetics, new biomarkers, risk factors of DR.

Objective:

1. To validate the methodology and feasibility of DR screening using a DL based automated DR grading system in clinical practice.
2. To explore the prevalence of DR and subgroup identification, and fundus images analysis, etc.
3. To explore the genetics, new biomarkers, risk factors of DR.
4. To explore the methods of early screening, prevention, treatment and referal process of DR.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for type 2 diabetes according to the World Health Organization (WHO) in 1999; Type 1 diabetes, single gene mutation diabetes, secondary diabetes caused by pancreatic damage, Cushing's syndrome, thyroid dysfunction, or acromegaly;
* Subjects from other medical institutes are diabetes, non-diabetic patients and healthy participants who are invited to participate in the study.

Exclusion Criteria:

* Those who have a history of drug abuse;
* Sexually transmitted diseases such as AIDS and syphilis, and infectious diseases such as viral hepatitis and tuberculosis which are at active phase;
* Any condition that the investigator think that the subject is not suitable for participating in the study.

For detailed In-/Ex-clusion criteria please see the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetes patients under the management of MMC, and diabetes, non-diabetic, and healthy participants from other medical institutes who meet the In-/Ex-clusion Criteria will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2038-06-05 (Estimated); Study Completion 2040-06-05 (Estimated)

PRIMARY OUTCOMES:
Diabetic retinopathy | through study completion, up to 20 years
  diabetic retinopathy
Referable diabetic retinopathy | through study completion, up to 20 years
  Referable diabetic retinopathy
Vision threatening diabetic retinopathy | through study completion, up to 20 years
  Vision threatening diabetic retinopathy
Diabetic macular edema | through study completion, up to 20 years
  Diabetic macular edema

SECONDARY OUTCOMES:
HbA1c (%) | through study completion, up to 20 years
Smoking history | through study completion, up to 20 years
Alcohol intake | through study completion, up to 20 years
Salt intake | through study completion, up to 20 years
Vegetable and fruits intake | through study completion, up to 20 years
Physical activity | through study completion, up to 20 years
Blood pressures (mmHg) | through study completion, up to 20 years
Lipids (mg/dl) | through study completion, up to 20 years
Cardiolvascular diseases | through study completion, up to 20 years
Body mass index (BMI) | through study completion, up to 20 years
  Body weight (kg) and height (m) will be combined to report BMI in kg/m^2
Systolic blood pressure | through study completion, up to 20 years
Diastolic blood pressure | through study completion, up to 20 years
Visceral fat (cm^2) | through study completion, up to 20 years
Fasting glucose (mmol/L) | through study completion, up to 20 years
Postprandial glucose (mmol/L) | through study completion, up to 20 years
Fasting serum C peptide (ug/L) | through study completion, up to 20 years
Postprandial serum C peptide (ug/L) | through study completion, up to 20 years
Fasting serum insuline (μIU/mL) | through study completion, up to 20 years
Postprandial serum insuline (μIU/mL) | through study completion, up to 20 years
Intimal medial thikness (mm) | through study completion, up to 20 years
Pulse wave velocity (cm/s) | through study completion, up to 20 years
Albumin-creatinine-ratio (mg/mmol) | through study completion, up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD,PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine Shanghai, Shanghai, China
Locations (2):
- China (2):
  - Ruijin hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Jiao-Tong University School of Medicine, Shanghai

REFERENCES:
- [Derived] Zhang Y, Shi J, Peng Y, Zhao Z, Zheng Q, Wang Z, Liu K, Jiao S, Qiu K, Zhou Z, Yan L, Zhao D, Jiang H, Dai Y, Su B, Gu P, Su H, Wan Q, Peng Y, Liu J, Hu L, Ke T, Chen L, Xu F, Dong Q, Terzopoulos D, Ning G, Xu X, Ding X, Wang W. Artificial intelligence-enabled screening for diabetic retinopathy: a real-world, multicenter and prospective study. BMJ Open Diabetes Res Care. 2020 Oct;8(1):e001596. doi: 10.1136/bmjdrc-2020-001596. PMID 33087340